CLINICAL TRIAL: NCT03518632
Title: Preoperative Physical Activity Intervention in Patients Before Planned Liver Resection for Cancer
Brief Title: Preoperative Physical Activity Intervention in Patients Before Planned Liver Resection for Cancer (APACHE)
Acronym: APACHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Célia Turco (Other)
Responsible Party: Sponsor-Investigator, Célia Turco, Principal Investigator, Centre Hospitalier Universitaire de Besancon
Organization: Centre Hospitalier Universitaire de Besancon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-A02992-51
Record Dates: First submitted 2018-04-06; First posted 2018-05-08 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2020-07

CONDITIONS: Primary Liver Cancer; Secondary Liver Cancer; Liver Metastases
Keywords: Exercise; Adapted physical activity; preoperative; liver resection; hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator)
  Interventions: Other: Standard Oncologic care
- Interval training 1 (Experimental)
  Interventions: Behavioral: Interval training
- Interval training 2 (Experimental)
  Interventions: Behavioral: Interval training

INTERVENTIONS:
Behavioral: Interval training — Patients in experimental group will perform a 6 weeks' physical activity program with 3 sessions per week. Physical activity intervention will consist in 2 different interval training programs on cycloergometer: Interval training 1 and Interval training 2, with a difference in exercise intensities.
  Arms: Interval training 1; Interval training 2
Other: Standard Oncologic care — Patients in control group will follow the standard oncologic care. They will perform only 2 sub-maximal exercises.
  Arms: Control group

SUMMARY:
The aim of this study is to assess the impact of preoperative physical activity on physical capacities of patients undergoing liver resection for primary or secondary liver cancer.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of a preoperative exercise program in patients with primary or secondary liver cancer undergoing hepatectomy. Preoperative exercise programs have been shown to be effective in other cancer populations, but have been poorly studied in patients with liver cancer. For these patients, it remains unclear what the optimal composition of such programs should be and how they should be delivered. Outcome measures in this study will include preoperative outcomes (oxygen consumption, quality of life, fatigue and physical activity level, anthropometric measures, plasma concentrations of hepatokines) and postoperative outcomes (length of hospital stay and postoperative complications).

After the study is explained and consent obtained, subjects will be tested on a submaximal exercise on cycloergometer with gas exchanges analysis and with pre and post blood test. Then, they will answer various questionnaires assessing physical activity, quality of life and fatigue.

Patients scheduled for liver resection will be randomized to one of two groups. The first group (experimental group) will be subdivided into two groups: interval training 1 and interval training 2, which differentiate themselves by two different intensities.The second group (control group) will receive standard care.

The prehabilitation program will last 6 weeks with 3 sessions per week and will consist in two interval training programs on a cycloergometer with two different intensities.

One month after surgery, peri and postoperative complications will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years old.
* Patients with primary liver cancer, biliary tract cancer, liver metastasis endorsed in the University Hospital of Besancon
* No opposition of patients
* Join a French social security or receiving such a scheme

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Patients being in the disqualification of another study or under the national register of volunteers
* Patients unlikely to cooperate or anticipated low cooperation
* Patients with a maximal oxygen consumption above 35 ml/min/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Oxgen consumption at anaerobic threshold : | 6 weeks
  Oxygen consumption at anaerobic threshold will be assessed at baseline and at the end of the 6 weeks' program with a submaximal exercise performed on cycloergometer

SECONDARY OUTCOMES:
Postoperative complications with the Dindo Clavien classification : | One month after surgery
  Postoperative complications will be assessed using the Dindo Clavien classification which consists in a 7 grades classification (I, II, IIIa, IIIb, IVa, IVb and V).
Intensive care stay : | One month after surgery
  Postoperative intensive care stay will be evaluated (number of days).
Changes of Hepatokines plasmatic concentrations : | Comparison between plasmatic concentrations pre-exercise (day 1), post exercise (day 1) and at 6 weeks
  Fetuin A (ng/mL) concentrations will be analyzed.
Hepatokines plasmatic concentrations : | Comparison between plasmatic concentrations pre-exercise (day 1), post exercise (day 1) and at 6 weeks
  Fibroblast Growth Factor 21 (FGF21) (pg/mL) concentrations will be analyzed.
Changes in Physical activity level : | Comparison between baseline, after the 6 weeks' program
  Physical activity level will be measured using the long-form of the International Physical Activity Questionnaire (IPAQ). It consist in a description of the physical activity level by assessing 5 activity domains during the 7 last days. Physical activity level is expressed in Metabolic Equivalent Tasks (METs). It enables to classify patients in 3 categories : low physical activity level, moderate physical activity level and high physical activity level.
Changes in Quality of life : | Comparison between baseline, after the 6 weeks' program
  Health related quality of life will be measured with the EORTC Quality of Life Questionnaire QLQ-C30 which is a cancer specific questionnaire. It consists in 30 items to measure 15 dimensions of quality of life. It generates a score between 0 and 100. A higher score means a higher quality of life level.
Changes in Fatigue : | Comparison between baseline, after the 6 weeks' program
  Fatigue will be measured with the Quality of Life Questionnaire QLQ-FA12 which enables to assess cancer related fatigue. It consists in 12 items to measure 5 dimension go health related fatigue. It generates a score between 0 and 100. A higher score means a higher fatigue level.

CONTACTS AND LOCATIONS:
Locations (1):
- Chirurgie digestive, viscérale et cancérologique, Besançon, France